CLINICAL TRIAL: NCT04571112
Title: Multi-targets, Single-lead GPi+NBM DBS in Parkinson's Disease With Mild Cognitive Impairment
Brief Title: GPi+NBM DBS in Parkinson's Disease With Mild Cognitive Impairment
Acronym: 2T-DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Dr. Alfonso Fasano, MD, PhD, Professor, Department of Medicine, Division of Neurology at University of Toronto, Toronto Western Hospital, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17-5400-B
Record Dates: First submitted 2019-09-12; First posted 2020-09-30 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease; Memory Disorders
MeSH Terms: conditions — Parkinson Disease; Memory Disorders

STUDY DESIGN:
Intervention Model Description: To target both the NBM and GPi in a single trajectory, using the Vercise system (Boston Scientific, Marlborough, Massachusetts, US) which is now approved for human use in Canada. This system includes a novel 8-contact electrode and an IPG system with 16 independent power sources allowing the so-called 'Multiple Independent Current Control' (MICC) that permits concurrent high- and low-frequency stimulation, as well as a variety of amplitudes and pulse widths independently controlled at each stimulated region.
Who Masked: Participant, Outcomes Assessor
Masking Description: * The post-surgical double-blind cross-over phase with randomization will follow once programming settings are determined. Under constant GPi DBS, patients will receive NBM DBS active or sham for 8 weeks followed by an 8-week cross-over. Then, patients will enter a post-surgical open-label follow-up phase during which they will receive GPi+NBM DBS.
  * The outcomes assessor is blinded to the whether the NBM DBS is active to avoid bias while analyzing the data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NBM ON (Experimental): The post-surgical double-blind cross-over phase with randomization will follow once programming settings are determined. Under constant GPi DBS, patients will receive NBM DBS active or sham for 8 weeks followed by an 8-week cross-over.
  The NBM ON arm will have constant NBM stimulation for 8 weeks.
  Interventions: Device: NBM stimulation using the Vercise device (Boston Scientific, Marlborough, Massachusetts, US)
- NBM OFF (Sham Comparator): The post-surgical double-blind cross-over phase with randomization will follow once programming settings are determined. Under constant GPi DBS, patients will receive NBM DBS active or sham for 8 weeks followed by an 8-week cross-over.
  The NBM OFF arm will have NBM stimulation turned off for 8 weeks.
  Interventions: Device: NBM stimulation using the Vercise device (Boston Scientific, Marlborough, Massachusetts, US)

INTERVENTIONS:
Device: NBM stimulation using the Vercise device (Boston Scientific, Marlborough, Massachusetts, US) — This will either be turned on or off depending on the arm which the patient is randomized to. After 8-weeks, the subject will switch arms for another 8-weeks.

SUMMARY:
This study examines the safety and feasibility of DBS in treating the movement and cognitive dysfunction in Parkinson's disease (PD). Globus pallidus interna (GPi) stimulation is an established treatment for the motor symptoms in PD, but it does not treat the cognitive symptoms that can also be seen in this condition. It is theorized that we can improve cognitive dysfunction by stimulating a part of the brain called the nucleus basalis of Meynert (NBM), which releases a chemical (acetylcholine) and plays a role in memory and attention. By using a novel DBS system (Vercise device) with 2 electrodes that are designed to stimulate the GPi and NBM, we can potentially target the motor and cognitive symptoms of PD with a single intervention.

DETAILED DESCRIPTION:
Neuronal loss within the cholinergic nucleus basalis of Meynert (NBM) correlates with cognitive decline in dementing disorders such as Alzheimer's disease and Parkinson's disease (PD). Deep Brain Stimulation targeting the Globus Pallidus interna (GPi) is an established treatment for the motor symptoms in Parkinson's Disease, and stimulating the NBM is believed to stimulate cognitive function. Targeting these two regions was previously impossible because they require different frequency stimulations, but recent developments in DBS technology allow for the dual stimulation of these nuclei at different frequencies.

This phase-II double-blind cross-over pilot trial will investigate the motor and cognitive effects as well as the presence of adverse effects of combined NBM and GPi DBS. The main goal of this pilot trial is to demonstrate the feasibility and safety of the multi-targeting approach in 6 patients with PDD and disabling motor symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. PD-MCI that affects multiple cognitive domains (including memory, visuo-spatial deficits etc.). diagnosis based on a comprehensive neuropsychological assessment (gold-standard) allowing the application of Level II MDS diagnostic criteria (Dubois et al. 2007)
2. PD fulfilling standard criteria for bilateral GPi DBS surgery
3. Patient's ability to provide informed consent and comply with study protocol.

Exclusion Criteria:

1. Severe Parkinson's disease dementia, preventing completion of the neuropsychological assessment, compliance with the study protocol, or ability to provide informed consent.
2. Inability to be fluent in English.
3. Unstable dose of any cognitive enhancing medication.
4. Presence of other neurological disorders, severe active psychiatric conditions or previous brain surgery.

Other conditions contraindicating DBS, PET scanning or MRI scanning.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in cognition after GPi/NBM DBS | at baseline and 6, 14, 22, 30 and 52 weeks post surgery
  This will be measured by the ADAS-Cog 13, verbal fluency test and sustained attention task.
Change in motor function (UPDRS)GPi/NBM DBS | at baseline and 6, 14, 22, 30 and 52 weeks post surgery
  Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a comprehensive 65 item assessment of both motor and non-motor symptoms associated with Parkinson's Disease. Each symptom is rated on a 5-point scale (from 0 to 4), and the maximum total score is 199, indicating severe impairment from parkinson's disease.
To assess the occurrence of adverse events from GPi/NBM DBS and occurrence of adverse events. | through study completion, an average of 1 year
  We define an adverse event (AE) as any untoward medical occurrence that occurs in the course of this study whether or not considered related to the study device, study procedures or study requirements that is identified or worsens during the study.

SECONDARY OUTCOMES:
To assess the impact on health-related quality-of-life and various non-motor symptoms of PD | 1 year
  This is measured by the Parkinson's Disease Questionnaire, with a score range from 0 (never have difficulty) to 100 (always have difficulty), and with lower scores reflecting a better quality of life
To use neuroimaging biomarkers (MEG and FDG-PET) to examine localized effects of NBM stimulation | with NBM turned on and off, 22 and 30 weeks after surgery respectively
  Region of interest analysis will be used to determine the localized effects of NBM in the surrounding structures and cortex for both MEG and PET imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Fasano, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bentley P, Driver J, Dolan RJ. Cholinergic modulation of cognition: insights from human pharmacological functional neuroimaging. Prog Neurobiol. 2011 Sep 1;94(4):360-88. doi: 10.1016/j.pneurobio.2011.06.002. Epub 2011 Jun 17. PMID 21708219
- [Background] Bosboom JL, Stoffers D, Stam CJ, Berendse HW, Wolters ECh. Cholinergic modulation of MEG resting-state oscillatory activity in Parkinson's disease related dementia. Clin Neurophysiol. 2009 May;120(5):910-5. doi: 10.1016/j.clinph.2009.03.004. Epub 2009 Apr 21. PMID 19386543
- [Background] Combs HL, Folley BS, Berry DT, Segerstrom SC, Han DY, Anderson-Mooney AJ, Walls BD, van Horne C. Cognition and Depression Following Deep Brain Stimulation of the Subthalamic Nucleus and Globus Pallidus Pars Internus in Parkinson's Disease: A Meta-Analysis. Neuropsychol Rev. 2015 Dec;25(4):439-54. doi: 10.1007/s11065-015-9302-0. Epub 2015 Oct 12. PMID 26459361
- [Background] Di Santo SG, Prinelli F, Adorni F, Caltagirone C, Musicco M. A meta-analysis of the efficacy of donepezil, rivastigmine, galantamine, and memantine in relation to severity of Alzheimer's disease. J Alzheimers Dis. 2013;35(2):349-61. doi: 10.3233/JAD-122140. PMID 23411693
- [Background] Dubois B, Burn D, Goetz C, Aarsland D, Brown RG, Broe GA, Dickson D, Duyckaerts C, Cummings J, Gauthier S, Korczyn A, Lees A, Levy R, Litvan I, Mizuno Y, McKeith IG, Olanow CW, Poewe W, Sampaio C, Tolosa E, Emre M. Diagnostic procedures for Parkinson's disease dementia: recommendations from the movement disorder society task force. Mov Disord. 2007 Dec;22(16):2314-24. doi: 10.1002/mds.21844. PMID 18098298
- [Background] Fasano A, Appel-Cresswell S, Jog M, Zurowkski M, Duff-Canning S, Cohn M, Picillo M, Honey CR, Panisset M, Munhoz RP. Medical Management of Parkinson's Disease after Initiation of Deep Brain Stimulation. Can J Neurol Sci. 2016 Sep;43(5):626-34. doi: 10.1017/cjn.2016.274. PMID 27670207
- [Background] Freund HJ, Kuhn J, Lenartz D, Mai JK, Schnell T, Klosterkoetter J, Sturm V. Cognitive functions in a patient with Parkinson-dementia syndrome undergoing deep brain stimulation. Arch Neurol. 2009 Jun;66(6):781-5. doi: 10.1001/archneurol.2009.102. PMID 19506141
- [Background] Gratwicke J, Jahanshahi M, Foltynie T. Parkinson's disease dementia: a neural networks perspective. Brain. 2015 Jun;138(Pt 6):1454-76. doi: 10.1093/brain/awv104. Epub 2015 Apr 16. PMID 25888551
- [Background] Kuhn J, Hardenacke K, Lenartz D, Gruendler T, Ullsperger M, Bartsch C, Mai JK, Zilles K, Bauer A, Matusch A, Schulz RJ, Noreik M, Buhrle CP, Maintz D, Woopen C, Haussermann P, Hellmich M, Klosterkotter J, Wiltfang J, Maarouf M, Freund HJ, Sturm V. Deep brain stimulation of the nucleus basalis of Meynert in Alzheimer's dementia. Mol Psychiatry. 2015 Mar;20(3):353-60. doi: 10.1038/mp.2014.32. Epub 2014 May 6. PMID 24798585
- [Background] Kumar R, Lang AE, Rodriguez-Oroz MC, Lozano AM, Limousin P, Pollak P, Benabid AL, Guridi J, Ramos E, van der Linden C, Vandewalle A, Caemaert J, Lannoo E, van den Abbeele D, Vingerhoets G, Wolters M, Obeso JA. Deep brain stimulation of the globus pallidus pars interna in advanced Parkinson's disease. Neurology. 2000;55(12 Suppl 6):S34-9. PMID 11188973
- [Background] Liu AK, Chang RC, Pearce RK, Gentleman SM. Nucleus basalis of Meynert revisited: anatomy, history and differential involvement in Alzheimer's and Parkinson's disease. Acta Neuropathol. 2015 Apr;129(4):527-40. doi: 10.1007/s00401-015-1392-5. Epub 2015 Jan 30. PMID 25633602
- [Background] McGaughy J, Kaiser T, Sarter M. Behavioral vigilance following infusions of 192 IgG-saporin into the basal forebrain: selectivity of the behavioral impairment and relation to cortical AChE-positive fiber density. Behav Neurosci. 1996 Apr;110(2):247-65. doi: 10.1037//0735-7044.110.2.247. PMID 8731052
- [Background] Mohs RC, Knopman D, Petersen RC, Ferris SH, Ernesto C, Grundman M, Sano M, Bieliauskas L, Geldmacher D, Clark C, Thal LJ. Development of cognitive instruments for use in clinical trials of antidementia drugs: additions to the Alzheimer's Disease Assessment Scale that broaden its scope. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S13-21. PMID 9236948
- [Background] Pagano G, Rengo G, Pasqualetti G, Femminella GD, Monzani F, Ferrara N, Tagliati M. Cholinesterase inhibitors for Parkinson's disease: a systematic review and meta-analysis. J Neurol Neurosurg Psychiatry. 2015 Jul;86(7):767-73. doi: 10.1136/jnnp-2014-308764. Epub 2014 Sep 15. PMID 25224676
- [Background] Park M, Hood MM, Shah RC, Fogg LF, Wyatt JK. Sleepiness, parkinsonian features and sustained attention in mild Alzheimer's disease. Age Ageing. 2012 Nov;41(6):765-70. doi: 10.1093/ageing/afs084. Epub 2012 Jun 27. PMID 22743151
- [Background] Picillo M, Lozano AM, Kou N, Puppi Munhoz R, Fasano A. Programming Deep Brain Stimulation for Parkinson's Disease: The Toronto Western Hospital Algorithms. Brain Stimul. 2016 May-Jun;9(3):425-437. doi: 10.1016/j.brs.2016.02.004. Epub 2016 Feb 12. PMID 26968806
- [Background] Ponce FA, Asaad WF, Foote KD, Anderson WS, Rees Cosgrove G, Baltuch GH, Beasley K, Reymers DE, Oh ES, Targum SD, Smith GS, Lyketsos CG, Lozano AM; ADvance Research Group. Bilateral deep brain stimulation of the fornix for Alzheimer's disease: surgical safety in the ADvance trial. J Neurosurg. 2016 Jul;125(1):75-84. doi: 10.3171/2015.6.JNS15716. Epub 2015 Dec 18. PMID 26684775
- [Background] Rolinski M, Fox C, Maidment I, McShane R. Cholinesterase inhibitors for dementia with Lewy bodies, Parkinson's disease dementia and cognitive impairment in Parkinson's disease. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD006504. doi: 10.1002/14651858.CD006504.pub2. PMID 22419314
- [Background] Rouaud T, Dondaine T, Drapier S, Haegelen C, Lallement F, Peron J, Raoul S, Sauleau P, Verin M. Pallidal stimulation in advanced Parkinson's patients with contraindications for subthalamic stimulation. Mov Disord. 2010 Sep 15;25(12):1839-46. doi: 10.1002/mds.23171. PMID 20568094
- [Background] Sarter M, Givens B, Bruno JP. The cognitive neuroscience of sustained attention: where top-down meets bottom-up. Brain Res Brain Res Rev. 2001 Apr;35(2):146-60. doi: 10.1016/s0165-0173(01)00044-3. PMID 11336780
- [Background] Smith GS, Laxton AW, Tang-Wai DF, McAndrews MP, Diaconescu AO, Workman CI, Lozano AM. Increased cerebral metabolism after 1 year of deep brain stimulation in Alzheimer disease. Arch Neurol. 2012 Sep;69(9):1141-8. doi: 10.1001/archneurol.2012.590. PMID 22566505
- [Background] Witt K, Daniels C, Krack P, Volkmann J, Pinsker MO, Kloss M, Tronnier V, Schnitzler A, Wojtecki L, Botzel K, Danek A, Hilker R, Sturm V, Kupsch A, Karner E, Deuschl G. Negative impact of borderline global cognitive scores on quality of life after subthalamic nucleus stimulation in Parkinson's disease. J Neurol Sci. 2011 Nov 15;310(1-2):261-6. doi: 10.1016/j.jns.2011.06.028. Epub 2011 Jul 5. PMID 21733529